CLINICAL TRIAL: NCT04088643
Title: The Efficacy of 4Hz Transcranial Alternating Current Stimulation for Patients With Mild Alzheimer's Disease: A Randomized Controlled Clinical Trial
Brief Title: 4Hz Transcranial Alternating Current Stimulation for Patients With Mild Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018077
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tACS group (Experimental): NEXALIN ADI transcranial alternating current stimulator
  Interventions: Device: transcranial alternating current stimulation
- sham stimulation group (Sham Comparator): Sham stimulator provided by NEXALIN company
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: transcranial alternating current stimulation — The alternating current is administered through medical grade conductive pads that are produced specifically for the Nexalin technology. The pads are places on the forehead and behind each ear, and are connected to the Nexalin device with thin cables. Intervention will be implemented with a tACS device with 4Hz frequency and a peak-to-peak amplitude of 15mA, 30 one-hour sessions in 3 weeks (21 days).
  Arms: tACS group
Device: sham stimulation — Electrodes will also be put on patient's forehead and behind each ear. The sham stimulator has the exactly same appearance with the true stimulator. Participants and operators cannot determine whether the stimulator is true based on its appearance or patients' feelings. However, when the device is started, no current flows through the electrodes. Participants in this controlled group will also receive sham stimulations with 30 one-hour sessions in 21 days.
  Arms: sham stimulation group

SUMMARY:
The goal of this study is to explore the efficacy and safety of 4Hz transcranial alternating current stimulation (tACS) in patients with mild Alzheimer's disease (AD). The study will recruit 40 individuals with mild AD, and the participants will be randomized to either a 4 Hz tACS group or a sham stimulation group. Both groups will undergo 30 one-hour sessions across 3 weeks (21 days). At the end of the intervention and 3-month follow-up, all subjects will repeat the baseline assessments.

DETAILED DESCRIPTION:
Background: Recently, transcranial alternating current stimulation (tACS), which could interact with ongoing neuronal activity, has emerged as a potentially effective and promising treatment for Alzheimer's disease (AD), and the 4Hz frequency was suggested to improve working memory Methods: The proposed study is a double-blinded, randomized controlled trial that will include 40 individuals with mild AD, and the participants will be randomized to either a 4Hz tACS group or a sham stimulation group. Both groups will undergo 30 one-hour sessions in 3 weeks (21 days). The outcome measures will be assessed at baseline, end of intervention and 3 months after the first session. Primary outcome is global cognitive function, assessed by the 11-item cognitive subscale of the Alzheimer's Disease Assessment Scale (ADAS-cog), and the second outcomes include changes in other neuropsychological assessments, structural MRI, resting electroencephalogram (EEG) and simultaneous EEG-functional MRI (fMRI).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with informed consent;
2. 45-75 years of age;
3. At least 6 years of education;
4. AD according to the National Institute on Aging and the Alzheimer's Association (NIA-AA) guidelines;
5. Clinical Dementia Rating Scale (CDR)=1.0;
6. Positive findings in amyloid PET imaging or amyloid protein levels in CSF;
7. On a stable dose of cholinesterase inhibitors (e.g. donepezil or rivastigmine) as defined as 6 consecutive weeks of treatment at an unchanging dose, and without any intentions to modify the dosage during the observation period.

Exclusion Criteria:

1. Current or past history of any neurological disorder other than dementia, such as epilepsy, stroke, progressive neurologic disease (e.g. multiple sclerosis), poorly controlled migraines or intracranial brain lesions; and history of previous neurosurgery or head trauma that resulted in residual neurologic impairment;
2. Contraindication for undergoing MRI or receiving tACS;
3. Eczema or sensitive skin;
4. Familial AD;
5. Depression or other psychiatric disorders;
6. Abnormal brain structural magnetic resonance imaging (MRI) scan, including hydrocephalus, stroke, structural lesions, etc. that would potentially confound the outcome;
7. Severe cardiovascular/pulmonary disorders;
8. Other conditions, in the investigator's opinion, might not be suitable for the study.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale cognitive subscale (ADAS-cog, 11-items version) | up to 21 days (end of intervention)
  ADAS-cog 11 scale ranges from 0 to 70, and higher value represents a worse outcome. This study will use ADAS-cog to assess changes in the global cognitive function after intervention.

SECONDARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale cognitive subscale (ADAS-cog, 11-items version). | 3 months
  ADAS-cog 11 scale ranges from 0 to 70, and higher value represents a worse outcome. This study will use ADAS-cog to assess changes in the global cognitive function after intervention.
Change in brain volume and white matter integrity | up to 21 days (end of intervention), 3 months
  Structural MRI will be used to measure brain volume and white matter integrity.
Change in brain connectivity | up to 21 days (end of intervention), 3 months
  Functional MRI and resting-state EEG will be used to measure brain connectivity.
Change in Mini-mental State Examination | up to 21 days (end of intervention), 3 months
  Mini-mental State Examination (MMSE) will be used to evaluate the general cognitive function. MMSE ranges from 0 to 30, and higher value represents a better outcome.
Change in Montreal Cognitive Assessment | up to 21 days (end of intervention), 3 months
  Montreal Cognitive Assessment (MoCA) will be used to evaluate the general cognitive function. MoCA ranges from 0 to 30, and higher value represents a better outcome.
Change in Clinical Dementia Rating Scale sum of the boxes | up to 21 days (end of intervention), 3 months
  Clinical Dementia Rating Scale sum of the boxes (CDR-SB) will be used to evaluate the general cognitive function. CDR-SB ranges from 0 to 18, and higher value represents a worse outcome.
Change in memory function | up to 21 days (end of intervention), 3 months
  WHO-UCLA Auditory Verbal Learning Test will be used to assess memory function. It ranges from 0 to 45, and higher value represents a better outcome.
Change in Digit span forward | up to 21 days (end of intervention), 3 months
  Digit span will be used to assess attention. It ranges from 3 to 10, and higher value represents a better outcome.
Change in Digit span backward | up to 21 days (end of intervention), 3 months
  Digit span backward will be used to assess executive function. It ranges from 2 to 8, and higher value represents a better outcome.
Change in Trail Making Test | up to 21 days (end of intervention), 3 months
  Trail-Making Test B minus A score will be used to assess executive function. Trail-Making Test B minus A ranges from -150 to 300, higher value represents a worse outcome.
Change in Boston Naming Test | up to 21 days (end of intervention), 3 months
  Boston Naming Test will be used to assess language function. It ranges from 0 to 30, and higher value represents a better outcome.
Change in Neuropsychiatric Inventory (NPI) | up to 21 days (end of intervention), 3 months
  The Neuropsychiatric Inventory will be used to measure neuropsychiatric symptoms. It ranges from 0 to 144, and higher value represents a worse outcome.
Change in Geriatric Depression Scale (GDS) | up to 21 days (end of intervention), 3 months
  The Geriatric Depression Scale will be used to measure neuropsychiatric symptoms. It ranges from 0 to 30, and higher value represents a worse outcome.
Change in Activities of Daily Living | up to 21 days (end of intervention), 3 months
  Activities of Daily Living (ADL) scale will be used to assess the change of life quality. It ranges from 20 to 80. The "20" represents normal life ability and the higher score presents the worse life ability.
Side-effects of tACS | up to 21 days (end of intervention), 3 months
  Adverse Events as a result of tACS stimulation will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Tang, M.D., Ph.D., Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China